CLINICAL TRIAL: NCT05630482
Title: Adaptation of an Evidence-based Family Program for Obesity Prevention in Health Care Context
Brief Title: Randomized Trial of Healthy Family Foundations
Acronym: HFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); State University of New York at Buffalo (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mark Feinberg, Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00020513; R01DK133525 (NIH)
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Family Foundations Intervention (Experimental): Participants randomized to the HFF intervention condition will participate in 10 weekly 2 hour classes (5 prenatal and 5 postnatal) in groups of 5-10 couples. Due to COVID, all classes will take place via Zoom. The classes will be led by male/female facilitator teams. The facilitators will be hired, trained and supervised by Penn State. Postnatal classes will occur 2-8 months after birth and will also be weekly and last 2 hours each.
  Interventions: Behavioral: Healthy Family Foundations
- Control Condition (Active Comparator): Participants randomized to the control condition will receive standard of care and opportunities for education at their site, including information about infant growth and development, infant care (including brief, standard information regarding breastfeeding/introduction to solid food), and quality childcare selection.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Healthy Family Foundations — Healthy Family Foundations Curriculum
  Arms: Healthy Family Foundations Intervention
Other: Standard of Care — Standard of Care
  Arms: Control Condition

SUMMARY:
The goal of this clinical trial is to test whether an adaptation of an evidence-based, couple-based preventive intervention at the transition to parenthood improves reduces obesity risk among infants and parents in military families via improved interparental support and coordination around health lifestyle behaviors and parenting.

The main question it aims to answer is whether an adapted, innovative family-focused approach to obesity prevention can reduce rapid infant weight gain, new mothers' postpartum weight retention, and fathers' weight status.

Participants randomized to the Healthy Family Foundations (HFF) intervention condition will participate in 10 online group classes (5 prenatal and 5 postnatal).

Participants randomized to the control condition will receive standard of care and opportunities for education at their site.

Researchers will compare the Healthy Family Foundations (HFF) intervention group with a Standard of Care control group to see if there are differences in weight, coparenting support, parent mental health and parent health behaviors.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test whether an adaptation of an evidence-based, couple-based preventive intervention at the transition to parenthood improves reduces obesity risk among infants and parents in military families via improved interparental support and coordination around health lifestyle behaviors and parenting.

The main question it aims to answer is whether an adapted, innovative family-focused approach to obesity prevention can reduce rapid infant weight gain, new mothers' postpartum weight retention, and fathers' weight status.

Aim 1. To assess the efficacy of the adapted HFF program with 275 military families from health centers at military bases in Washington, Florida, and Nevada. Families with an active-duty servicemember parent will be randomized to Healthy Family Foundations (HFF) or control condition. Primary outcomes consist of infant weight status (weight-for-length z-score) and maternal postpartum weight retention through 12 months; fathers' change in weight to 12 months is a secondary outcome.

Aim 2. To test mediation: HFF will foster healthy (A) parent weight outcomes via mutual parental support around healthy lifestyle behaviors (physical activity, nutrition, sleep); and (B) child weight status via coparenting support for health-related parenting (responsive feeding and promotion of sleep, physical activity, stress regulation).

Aim 3. To assess whether baseline parent characteristics (financial stress, mental health, relationship conflict, or weight status) or participant program engagement moderate program effects.

Participants randomized to the Healthy Family Foundations (HFF) intervention condition will participate in 10 online group classes (5 prenatal and 5 postnatal).

Participants randomized to the control condition will receive standard of care and opportunities for education at their site.

Researchers will compare the Healthy Family Foundations (HFF) intervention group with a Standard of Care control group to see if there are differences in weight, coparenting support, parent mental health and parent health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Two-parent military families (one or more parents are active duty military)
* Expecting a first child, through 7 months gestation

Exclusion Criteria:

* Clinical exclusion criteria for parents apply to males and females (active diagnosis of cancer, AIDS, palliative medicine patients, malabsorptive conditions, uncontrolled multiple sclerosis, and severe cognitive impairment), and to females (multiple gestation)
* Families will be excluded if both parents do not participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 825 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
BMI | 1 year
  weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale Revised (CESD-R-20) | 1 year
  The Center for Epidemiologic Studies Depression Scale (CESD). Scores range from 0-60, with higher scores indicating more depressive symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Feinberg, PhD, Principal Investigator — Penn State University
Locations (1):
- Nellis Airforce Base, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No